CLINICAL TRIAL: NCT03760237
Title: Cardiovascular Function in Leukemia Patients: an Observational Prospective Study
Brief Title: Cardiovascular Function in Acute Leukemia
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC48418
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-05

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphoid, Acute; Cardiotoxicity
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute Leukemia: Observation only. Patients newly diagnosed with acute leukemia who are scheduled to start treatment with chemotherapy will be enrolled and followed serially with blood collection, echocardiogram, arterial applanation tonometry, and questionnaires for 1 year.
  Interventions: Other: observation only

INTERVENTIONS:
Other: observation only — No intervention, observational study only

SUMMARY:
An observational, prospective study to describe the rates and predictors of cardiovascular events in patients with acute leukemia.

DETAILED DESCRIPTION:
Patients recently diagnosed with acute leukemia and who will initiating chemotherapy will be enrolled and followed serially with blood collection, echocardiogram, arterial applanation tonometry, and questionnaires for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age,
* New diagnosis of untreated acute leukemia (prior treatment for myelodysplastic syndrome or myeloproliferative neoplams or prior treatment with an anthracycline for breast cancer, Hodgkin's lymphoma, non-Hodgkin's lymphoma or another diagnosis will be included).
* Signed the informed consent form

Exclusion Criteria:

• Unable to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are newly diagnosed with acute leukemia
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Left Ventricular dysfunction | 1 year
  defined as a reduction in Left Ventricular Ejection Fraction of more than 10 percentage points from baseline and to less than 50%.

SECONDARY OUTCOMES:
Incidence of Cardiovascular Events | 1 year
Incidence of Symptomatic Heart Failure | 1 year
Incidence of Cardiac Death and all mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Scherrer-Crosbie, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided